CLINICAL TRIAL: NCT03263702
Title: Real-time Electrogram Analysis for Drivers of AtRial Fibrillation (RADAR)
Brief Title: RADAR Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Collaborators: AFTx, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 17-1537
Record Dates: First submitted 2017-06-28; First posted 2017-08-28 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Computational Mapping Algorithm (Experimental): AF mapping (utilizing CMA) will be performed and used to point the operator to regions within a heart chamber that should be interrogated further for suspicious electrogram activity, as measured by the St. Jude Ensite System, and ablated if the suspicious electrogram activity persists.
  Interventions: Device: Computational Mapping Algorithm

INTERVENTIONS:
Device: Computational Mapping Algorithm — This software enables high resolution temporospatial mapping of atria for the identification of drivers of AF. CMA receives data from standard of care, commercially available 3D Mapping Systems (St. Jude Ensite System) and catheters and processes the data in a unique way. Electrogram and anatomy data are fed from the commercially available 3D Mapping System to an adjacent laptop computer, via an Ethernet connection, that is running CMA. CMA then processes the electrogram data and generates a map of where the potential AF driver domains are located and superimposes those potential AF driver domain targets onto the 3D geometry of the anatomy (provided by the 3D mapping system).

SUMMARY:
This prospective, multicenter, observational study will examine the ability of real time electrogram processing mapping to identify driver domains to target for ablation in persistent AF patients.

DETAILED DESCRIPTION:
ABSTRACT: Recent clinical trials have shown that targeting rotors and focal impulses (FIs) during atrial fibrillation (AF) ablation improves outcomes. This study evaluated whether a novel computational mapping algorithm (CMA) could identify FIs and rotors, and characterize rotors when incidental ablation resulted in rhythm changes. Three-dimensional (3D) left atrial electroanatomic maps were created from signals recorded from multipolar circular mapping catheters in 61 patients undergoing persistent AF ablation. Forty of 61acquired patient datasets were of adequate quality for analysis CMA, employing an AF pattern recognition algorithm, creating 3D panoramic AF maps identifying drivers of AF (FI and rotors) post procedure. Rotors were further classified as substrate (SBR) or non-substrate based (NSBR) on the basis of rotor stability, proximity to voltage transition zones and complex fractionated atrial electrograms (CFAEs). Incidentally ablated identified AF drivers, including SBRs and NSBRs, were evaluated for rhythm changes. A total of 172 drivers were identified in 40 patients (2.2 drivers/patient). Seventy percent were rotors (120/172) and 30% were FIs (52/172). Sixty-seven percent of rotors were classified as SBR vs 33% as NSBR. Incidental ablation of SBRs resulted in rhythm change 91% of the time versus only 24% of the time for NSBR (p<0.0001).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Patients are considered eligible if they have symptomatic or drug-refractory AF and are planned to undergo a catheter ablation procedure for persistent AF (ether a first procedure or a redo procedure)
* Ability to understand the requirements of the study and sign the informed consent form.
* Willingness to adhere to study restrictions and comply with all post-procedural follow-up requirements
* Projected lifespan greater than 1 year.

Exclusion Criteria:

* They have long-standing persistent AF prior to the first procedure (defined as AF greater than one year's duration).
* Rheumatic heart disease
* Current intra-cardiac thrombus
* History of MI or Coronary Artery Bypass Grafting (CABG) within 6 weeks
* Unstable angina
* CVA or TIA within 3 months
* Contraindication to anticoagulation
* Class IV HF
* Unable to sign consent
* Projected lifespan of < 1 year
* Women known to be pregnant or to have positive beta-HCG (Human Chorionic Gonadotropin).
* Participation in another study that would interfere with this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - University of Colorado Medical Center, Denver, Colorado
  - South Denver Cardiology, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choudry S, Mansour M, Sundaram S, Nguyen DT, Dukkipati SR, Whang W, Kessman P, Reddy VY. RADAR: A Multicenter Food and Drug Administration Investigational Device Exemption Clinical Trial of Persistent Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2020 Jan;13(1):e007825. doi: 10.1161/CIRCEP.119.007825. Epub 2020 Jan 16. PMID 31944826

RESULTS

PARTICIPANT FLOW:
Groups:
- De Novo: Participants with 1st procedure
- Re-Do Ablation: Participants who need a re-do ablation procedure
Period: Overall Study
Arm/Group | De Novo | Re-Do Ablation
Started | 38 | 26
Completed | 35 | 22
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | De Novo | Re-Do Ablation | Total
Number analyzed (Participants) | 38 | 26 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.4) | 65.4 (9.9) | 64.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 26 | 21 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 37 | 25 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 36 | 24 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Atrial Fibrillation Termination
Description: Acute Procedural Outcomes as defined by termination of Atrial Fibrillation into normal sinus rhythm (NSR) or atrial tachycardia (AT)
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
Participants | 23 | 12

2. Primary Outcome: Number of Participants Free From Recurrent AT/AF on no AAD
Description: Number of Participants freedom from recurrent Atrial Tachycardia/Atrial Fibrillation with no use of Anti-Arrhythmic Drugs (AAD)
Time Frame: at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
Participants | 25 | 13

3. Primary Outcome: Number of Participants Free From Recurrent AT/AF With no or Some AAD
Description: Number of Participants Free recurrent Atrial Tachycardia/Atrial Fibrillation with either some or no use of Anti-Arrhythmic Drugs
Time Frame: at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
Participants | 25 | 17

4. Secondary Outcome: Rate of Post-ablation Inducibility of AF
Description: Post-ablation inducibility of AF (> 5 mins) with burst pacing
Time Frame: Day 1
Measure: Number; unit: percent of occurences
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
percent of occurences | 61 | 46

5. Secondary Outcome: Duration of RF Ablation
Description: Amount of radiofrequency ablation used for atrial fibrillation ablation
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
minutes | 323 (141.5) | 316 (88.56)

6. Secondary Outcome: Duration of Fluoro Time
Description: Duration of fluoroscopy used during the AF ablation procedure
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
minutes | 25.5 (13.1) | 24.1 (9.0)

7. Secondary Outcome: Duration of Exposure
Description: Radiation exposure due to fluoroscopy during the AF ablation procedure
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
mGy | 245 (201) | 241 (197)

8. Secondary Outcome: Duration of Procedure Time
Description: Duration of RADAR procedure time
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
minutes | 23.6 (20.3) | 34.5 (19.3)

9. Secondary Outcome: Number of Procedure-related Adverse Events
Time Frame: up to 12 months
Measure: Number; unit: events
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
events | 7 | 4

10. Secondary Outcome: Number of Major Adverse Cardiac Events (MACE)
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
events | 1 | 1

11. Secondary Outcome: Number of Serious Adverse Events
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | De Novo | Re-Do Ablation
Number analyzed (Participants) | 38 | 26
events | 12 | 8

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | De Novo | Re-Do Ablation
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/26
Serious Adverse Events (participants affected / at risk) | 10/38 | 5/26
Other Adverse Events (participants affected / at risk) | 8/38 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo (N=38) | Re-Do Ablation (N=26)
Amiodarone induced ataxia (Nervous system disorders) | 1 | 0
Amiodarone Intolerance (General disorders) | 1 | 0
Blood in stool (Gastrointestinal disorders) | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — lung infection
Cellulitis with lower back abscess (Skin and subcutaneous tissue disorders) | 0 | 1
COPD Exacebation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fever (Infections and infestations) | 1 | 0
Gastroesophageal bleed with hypotension (Gastrointestinal disorders) | 1 | 0
Generalized Weakness (General disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Non-sustained Ventricular Tachycardia (Cardiac disorders) | 2 | 0
Prostatectomy (Renal and urinary disorders) | 0 | 1
Pseudoaneurysm of right femoral artery (Vascular disorders) | 0 | 1 — with retroperitoneal hemorrhage
Severe Mitral Valve Regurgitation, and Paroxysmal Atrial Fibrillation (Cardiac disorders) | 1 | 0
Severe three vessel coronary artery disease (Cardiac disorders) | 1 | 0
Shortness of breath and abdominal rash (General disorders) | 0 | 1
Upper GI bleed (Gastrointestinal disorders) | 1 | 1
Worsening heart failure with influenza (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo (N=38) | Re-Do Ablation (N=26)
Chest pain (Cardiac disorders) | 0 | 1
Cogitive Decline (Nervous system disorders) | 1 | 0
Congestive Heart Failure (Cardiac disorders) | 1 | 0
Atypical flutter with RVR (Cardiac disorders) | 1 | 0
Fever (Infections and infestations) | 1 | 0
Fluid Overload (Cardiac disorders) | 1 | 0
Hematochezia (Gastrointestinal disorders) | 1 | 0
Lower extremity edema (Vascular disorders) | 1 | 0 — lower extremity edema with dyspnea and subsequent hypokalemia with diuresis
Pericarditis (Cardiac disorders) | 0 | 1
Peripheral Edema (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Recurrent Left Pleural Effusions (Cardiac disorders) | 1 | 0
Symptomatic PVCs (Cardiac disorders) | 1 | 1
Vaginitis (Renal and urinary disorders) | 1 | 0
Vertigo (Labyrinthitis) (General disorders) | 0 | 1
VF with ICD Shock (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT03263702/Prot_SAP_000.pdf